CLINICAL TRIAL: NCT05550116
Title: Clinical Evaluation of White Spot Lesions Treated by S-PRG Coating Material and Resin Sealants in Comparison With Resin Infiltration by Using Spectrophotometer and Laser Fluorescence. (A Randomized Controlled Trial) (WSLs)
Brief Title: Clinical Evaluation of White Spot Lesions Treated by S-PRG and ICON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Wakwak, Assistant professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2286488
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: White Spot Lesion
Keywords: white spot lesions; ICON; S-PRG; DIAGNOdent
MeSH Terms: interventions — PRG Barrier Coat; PermaSeal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Icon resin infiltration material (Active Comparator): Smooth surface resin infiltration comprises three steps for resin infiltration; Icon etch, Icon dry, and Icon infiltrant
  Interventions: Other: Giomer; Other: Two composite resin sealants
- PRG Barrier Coat (Experimental): fluoride-releasing coating material containing surface reaction-type pre-reacted glass-ionomer (S-PRG) fillers
  Interventions: Other: Two composite resin sealants
- Permaseal composite resin sealant (Experimental): Permaseal unfilled composite resin sealants
  Interventions: Other: Giomer
- Optiguard (Experimental): Optiguard unfilled composite resin sealant
  Interventions: Other: Giomer

INTERVENTIONS:
Other: Giomer — fluoride-releasing coating material containing surface reaction-type pre-reacted glass-ionomer (S-PRG) fillers
  Other Names: PRG Barrier Coat
  Arms: Icon resin infiltration material; Optiguard; Permaseal composite resin sealant
Other: Two composite resin sealants — Unfilled composite resin sealants
  Other Names: Permaseal and Optiguard
  Arms: Icon resin infiltration material; PRG Barrier Coat

SUMMARY:
Randomized with (1:1) prospective, double-blind, controlled trial. Subjects will be randomized to receive S-PRG and the control group receives ICON.

DETAILED DESCRIPTION:
Interventions: - All the procedures will be performed by the same clinician. DIAGNOdent will be used to assess the fluorescence loss of WSLs and the adjacent sound enamel. WSLs in permanent teeth will be treated according to the manufacturer's instructions with:

* Group I (Control group): 20 teeth will be treated with ICON.
* Group II ( EXPERIMENTAL) : 20 teeth will be treated with PRG BarrierCoat.

Observation: - The treatment methods will be assessed immediately after the intervention, 3 months,6 months, and one year. The data will be collected for evaluation of the difference in color and fluorescence loss between the treatment groups, by using DIAGNOdent devices, over different time intervals.

Ethical considerations: The research protocol is approved by the ethical committee, Faculty of Dental Medicine, Al-Azhar University and the enrolled patients should sign a written consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 20-40 years of age.
* Each patient has 4 or more WSLs.
* Mild and moderate WSLs according to Gorelick's scale.
* Good oral hygiene and willing patients who can attend the study visits.
* a Symmetrical number of permanent teeth in each arch (mesial to second molars).

Exclusion Criteria:

* Active carious lesions.
* Facial surface restorations.
* Intrinsic and extrinsic stains.
* Patients who have a significant medical history or if they smoke.
* Criteria for discontinuation; Mortality and acquiring severe debilitating disease

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-11 (Estimated)

PRIMARY OUTCOMES:
patients tooth color change | 1 year
  Color change with Vita Easyshade When the Delta E increased, it consider esthetic improving

SECONDARY OUTCOMES:
patients tooth caries lesion state | 1 year
  Laser fluorescence score Assessing of carious lesions state of the lesions by Diagnodent Minimum score is 0, while maximum score is 20 When score is decreased it consider positive results

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Noman, PROF, Study Director — Alazhar Univerisity
Locations (1):
- Mohamed Wakwak, Cairo, Egypt